CLINICAL TRIAL: NCT00887991
Title: Randomised Trial Comparing the Efficacy of the ISIS Duo iQ Electric Breast Pump and the Medela Symphony Electric Breast Pump in Mothers Expressing Breast Milk for Preterm Infants
Brief Title: A Trial Comparing Two Breast Pumps in Mothers Expressing Milk for Their Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Child Health (Other)
Responsible Party: Dr Mary Fewtrell, Institute of Child Health
Other Study IDs: 09NT02
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2009-04-24 (Estimated); Status verified 2009-04

CONDITIONS: Milk Production
Keywords: Randomised trial; breast pumps; efficacy; preterm; Mothers of preterm infants who plan to express milk for their infants.
MeSH Terms: conditions — Breast Milk Expression; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Electric Pump 1 (ISIS Duo iQ Electric Breast Pump): This is a parallel trial where subjects (mother of preterm infants) will be allocated to use one of two electric breast pumps to express milk. The use of electric breast pumps is routine practice on neonatal units in the UK.
- Electric Pump 2 (Medela Symphony Electric Breast Pump): This is a parallel trial where subjects (mother of preterm infants) will be allocated to use one of two electric breast pumps to express milk. The use of electric breast pumps is routine practice on neonatal units in the UK.

SUMMARY:
This is a randomised controlled trial investigating the performance of two, 'state of the art' electric breast pumps in mothers who have delivered preterm infants. The main data collection period will be up to day 10 post delivery data. Data collected will include a record of the weight of milk produced during the first 10 days and a short questionnaire to find the mothers' opinions of the pumps used. On Day 5 a timed and weighed expression of 15 minutes will be carried out. After the first 10 days, mothers will be asked to collect brief information on their continuing use of their pumps and subsequent duration of breast and bottle feeding, mothers will be contacted at 3 and 6 months post-term

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have delivered, preterm (before 34 weeks) infants who plan to express breast milk for their infant(s). Their infants will need to be less than 72 hours old prior to enrolment and likely to remain in NICUs for at least 10 days.

Exclusion Criteria:

* Other mothers not fitting inclusion criteria.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a parallel trial where subjects (mother of preterm infants) will be allocated to use one of two electric breast pumps to express milk.
Sampling Method: Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-07 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Total weight of milk expressed during the first 10 days post-partum. | 10 days post-partum
Weight of milk collected at 1 minute intervals over a 15 minute period on Day 5. | 10 days post-partum
Time taken to express a fixed volume of milk. | 10 days post-partum
Time taken for first milk to appear. | 10 days post-partum

SECONDARY OUTCOMES:
Total number of pumping sessions to Day 10. | 10 days
Total time spent expressing to Day 10. | 10 days
Mothers' opinions of the assigned pumps on Day 10. | 1 day
Volume of milk expressed whilst on neonatal unit. | 10 days
Number of days taken to reach full enteral feeds. | 10 or more days

CONTACTS AND LOCATIONS:
Overall Officials: Mary Fewtrell, Dr, Principal Investigator — Institute of Child Health; Pat Burton, Study Director — Institute of Child Health
Locations (1):
- Institute of Child Health, 30 Guilford Street, London, United Kingdom

REFERENCES:
- [Background] Fewtrell MS, Lucas P, Collier S, Singhal A, Ahluwalia JS, Lucas A. Randomized trial comparing the efficacy of a novel manual breast pump with a standard electric breast pump in mothers who delivered preterm infants. Pediatrics. 2001 Jun;107(6):1291-7. doi: 10.1542/peds.107.6.1291. PMID 11389245
- [Derived] Fewtrell MS, Kennedy K, Ahluwalia JS, Nicholl R, Lucas A, Burton P. Predictors of expressed breast milk volume in mothers expressing milk for their preterm infant. Arch Dis Child Fetal Neonatal Ed. 2016 Nov;101(6):F502-F506. doi: 10.1136/archdischild-2015-308321. Epub 2016 Mar 2. PMID 26936878
- [Derived] Burton P, Kennedy K, Ahluwalia JS, Nicholl R, Lucas A, Fewtrell MS. Randomized trial comparing the effectiveness of 2 electric breast pumps in the NICU. J Hum Lact. 2013 Aug;29(3):412-9. doi: 10.1177/0890334413490995. Epub 2013 Jun 17. PMID 23776081